CLINICAL TRIAL: NCT04398680
Title: A Phase I Study to Evaluate the Pharmacokinetics and Safety of Belantamab Mafodotin Monotherapy in Participants With Relapsed or Refractory Multiple Myeloma Who Have Normal and Varying Degrees of Impaired Hepatic Function (DREAMM 13)
Brief Title: A Study of Belantamab Mafodotin in Multiple Myeloma Participants With Normal and Impaired Hepatic Function
Acronym: DREAMM 13
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Sponsor Decision
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 209627
Expanded Access: NCT03763370 (Available)
Record Dates: First submitted 2020-05-19; First posted 2020-05-21 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-11

CONDITIONS: Multiple Myeloma
Keywords: DREAMM 13; Belantamab mafodotin monotherapy; Hepatic impairment; Normal hepatic function; Relapsed or refractory multiple myeloma
MeSH Terms: conditions — Multiple Myeloma; Recurrence | interventions — belantamab mafodotin

STUDY DESIGN:
Masking Description: This is an open-label study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Part 1, Group 1: Participants with normal hepatic function (Experimental): Participants with normal hepatic function (Serum bilirubin and Aspartate aminotransferase [AST] less than or equal to [<=] Upper limit of normal [ULN]) will be administered with Belantamab mafodotin
  Interventions: Drug: Belantamab mafodotin
- Part 1, Group 2: Participants with moderate hepatic impairment (Experimental): Participants with moderate hepatic impairment (Serum bilirubin greater than >1.5 - 3 times ULN and any AST) will be administered with Belantamab mafodotin
  Interventions: Drug: Belantamab mafodotin
- Part 2,Group 3: Participants with severe hepatic impairment (Experimental): Participants with severe hepatic impairment (Serum bilirubin >3 times ULN and any AST) will be administered with Belantamab mafodotin
  Interventions: Drug: Belantamab mafodotin

INTERVENTIONS:
Drug: Belantamab mafodotin — Belantamab mafodotin will be administered

SUMMARY:
The purpose of this study is to assess the pharmacokinetics (PK), safety, and tolerability of belantamab mafodotin monotherapy in Relapsed/Refractory Multiple Myeloma (RRMM) participants with impaired hepatic function and in matched RRMM participants with normal hepatic function.

ELIGIBILITY:
Inclusion Criteria:

* Participants are capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the Informed Consent Form.
* Male and/or female must be 18 years of age or older, at the time of signing the informed consent.
* Eastern Cooperative Oncology Group performance status 0-2.
* Participants with histologically or cytologically confirmed diagnosis of multiple myeloma, as defined in International Myeloma Working Group criteria: Has failed at least 1 prior line of anti-myeloma
* Participants has measurable disease with at least one of the following: Serum M-protein greater than or equal to (>=)0.5 grams per deciliter (g/dL) >=5 grams per liter [g/L]); Urine M-protein >=200 milligram per 24 hours (mg/24 hr); and Serum free light chain assay: Involved free light chain level >=10 milligrams per deciliter (mg/dL) (>=100 milligrams per liter [mg/L]); abnormal serum free light chain ratio (<0.26 or >1.65); participants with plasmacytoma and otherwise non-measurable disease
* Participants with a history of autologous SCT are eligible for study participation provided the following eligibility criteria are met: 1. Transplant was >100 days prior to study enrollment, 2. No active infection(s), and 3. Participant meets the remainder of the eligibility criteria outlined in this protocol.
* Participants with adequate organ system functions as defined below: Absolute neutrophil count >=1.0 times 10^9/liter (L); Hemoglobin >=8.0 g/dL (or 4.9 millimoles per liter); Platelets >= 75 times 10^9/L; Serum bilirubin and aspartate aminotransferase: Group 1 (normal) serum bilirubin and aspartate aminotransferase <=upper limit of normal (ULN); Group 2 (moderate) serum bilirubin >1.5-3 times ULN and any aspartate aminotransferase; alanine aminotransferase <=5 ULN; Estimated glomerular filtration rate >=30 milliliter per minute per 1.73 meter square (mL/min/m^2); Urine dipstick for protein or Albumin/creatinine ratio (from spot urine) negative/trace (if >=1+ only eligible if confirmed <=500 mg/g (56 mg/mmol) by albumin/creatinine ratio (spot urine from first void; and left ventricular ejection fraction by echocardiograms >=45 percent (%).
* Main additional inclusion criteria in Group 1 (matched control participants): Matched to at least one moderate hepatic impaired participant by Baseline albumin levels (+/-10%) and Baseline weight (+/-20%).
* Female participants: Contraceptive use by women should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies. A female participant is eligible to participate if she is not pregnant or breastfeeding, and not a woman of childbearing potential (WOCBP) or is a WOCBP and using a contraceptive method that is highly effective (with a failure rate of <1% per year).
* Male participants: Contraceptive use by men should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies. Male participants are eligible to participate if they agree to the following from the time of first dose of study until 6 months after the last dose of study treatment.
* Participants with a history of Hepatitis B virus and/or Hepatitis C virus and HIV exposure are eligible under specific conditions.

Exclusion Criteria:

* Active plasma cell leukemia at the time of screening. symptomatic amyloidosis, active polyneuropathy, organomegaly, endocrinopathy, myeloma protein and skin changes, Waldenstroem macroglobulinemia.
* Participants had a prior allogeneic SCT.
* Prior belantamab mafodotin therapy if given within the last 90 days.
* Systemic active infection requiring treatment
* Any unresolved toxicity >=Grade 2 from previous treatment except for alopecia, or peripheral neuropathy up to Grade 2.
* Any serious and/or unstable pre-existing medical, psychiatric disorder or other conditions (including lab abnormalities except hepatic impairment) that could interfere with participant's safety, obtaining informed consent or compliance to the study procedures.
* Current unstable liver or biliary disease per investigator assessment defined by the sudden onset of, or clinically relevant changes in: ascites, encephalopathy, coagulopathy, hypoalbuminemia, esophageal or gastric varices, persistent jaundice, in the last 14 days prior to the first dose.
* Participants with Hepatitis B will be excluded unless the following criteria can be met: If the participant is hepatitis B core antibody (HbcAb) positive or hepatitis B surface antigen (HbsAg) negative, then hepatitis B virus (HBV) deoxyribonucleic acid (DNA) should be undetectable at the time of screening; If HbsAg+ at screening or <=3 months prior to first dose of study treatment, then HBV DNA should be undetectable, highly effective antiviral treatment should be started ≥4 weeks prior to first dose of study treatment. Participants with cirrhosis are excluded.
* Positive hepatitis C antibody test result or positive hepatitis C ribonucleic acid test result at Screening or within 3 months prior to first dose of study treatment unless the participant can meet the following criteria: RNA test negative and/or Successful anti-viral treatment (usually 8 weeks duration) is required, followed by a negative HCV RNA test after a washout period of at least 4 weeks prior to first dose.
* Participants with Gilbert's syndrome.
* -Participants with previous or concurrent invasive malignancies other than MM are excluded, unless the prior malignancy has been considered medically stable for at least 1 year. The participant must not be receiving active therapy, other than hormonal therapy for this disease.
* Evidence of cardiovascular risk including any of the following: Evidence of current clinically significant untreated arrhythmias, including clinically significant electrocardiogram abnormalities including second degree (Mobitz Type II) or third degree atrioventricular block; History of myocardial infarction, acute coronary syndromes (including unstable angina), coronary angioplasty, or stenting or bypass grafting within 3 months of Screening; Class III or IV heart failure as defined by the New York Heart Association functional classification system; and Uncontrolled hypertension.
* Known human immunodeficiency virus infection, unless the participant can meet all of the following criteria: Established anti-retroviral therapy (ART) for at least 4 weeks and HIV viral load <400 copies/mL prior to first dose; CD4+ T-cell (CD4+) counts ≥350 cells/ L and no history of AIDS-defining opportunistic infections within the last 12 months.
* Current corneal epithelial disease except for mild punctuate keratopathy.
* Participant is a woman who is pregnant or breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-04-20 (Actual); Primary Completion 2025-11-04 (Estimated); Study Completion 2025-11-04 (Estimated)

PRIMARY OUTCOMES:
Part 1 and Part 2: Maximum observed plasma concentration (Cmax) of Belantamab Mafodotin | Up to 48 months
Part 1 and Part 2: Time to Cmax (Tmax) of Belantamab Mafodotin | Up to 48 months
Part 1 and Part 2: Concentration at the end of infusion (C-EOI) | Up to 48 months
Part 1 and Part 2: Predose plasma concentration (Ctrough) of Belantamab Mafodotin | Up to 48 months
Part 1 and Part 2: Area under the plasma concentration-time curve (from zero to the end of dosing interval) | Up to 48 months
Part 1 and Part 2: Last time point where the concentration is above the limit of quantification (Tlast) of Belantamab Mafodotin | Up to 48 months
Part 1 and Part 2: Cmax of total monoclonal antibody (mAb) | Up to 48 months
Part 1 and Part 2: Tmax of total mAb | Up to 48 months
Part 1 and Part 2: C-EOI of total mAB | Up to 48 months
Part 1 and Part 2: Ctrough of total mAb | Up to 48 months
Part 1 and Part 2: Area under the plasma concentration-time curve (from zero to the end of dosing interval)of total mAb | Up to 48 months
Part 1 and Part 2: Tlast of total mAb | Up to 48 months
Part 1 and Part 2: Cmax of Cys Monomethyl Auristatin F (cys-mcMMAF) | Up to 48 months
Part 1 and Part 2: Tmax of cys-mcMMAF | Up to 48 months
Part 1 and Part 2: C-EOI of cys-mcMMAF | Up to 48 months
Part 1 and Part 2: AUC(0-168 hours) of cys-mcMMAF | Up to 48 months
Part 1 and Part 2: tlast of cys-mcMMAF | Up to 48 months

SECONDARY OUTCOMES:
Part 1 and Part 2: Change from Baseline in Vital Signs- Diastolic Blood Pressure (DBP) and Systolic Blood Pressure (SBP) (millimeters of mercury [mmHg]) | Baseline and up to 4 years
Part 1 and Part 2: Change from Baseline in Vital Sign- Heart rate (beats per minute) | Baseline and up to 4 years
Part 1 and Part 2: Number of participants with adverse events (AEs) and serious adverse events (SAEs) | Up to 4 years
Part 1 and Part 2: Number of participants with toxicity grading for hematology parameters | Up to 4 years
Part 1 and Part 2: Number of participants with toxicity grading for clinical chemistry parameters | Up to 4 years
Part 1 and Part 2: Number of participants with toxicity grading for urine parameters | Up to 4 years

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (16):
- United States (8):
  - GSK Investigational Site, Tucson, Arizona
  - GSK Investigational Site, Beverly Hills, California
  - GSK Investigational Site, Plantation, Florida
  - GSK Investigational Site, Wichita, Kansas
  - GSK Investigational Site, Baltimore, Maryland
  - GSK Investigational Site, Monroeville, Pennsylvania
  - GSK Investigational Site, The Woodlands, Texas
  - GSK Investigational Site, Milwaukee, Wisconsin
- GSK Investigational Site, Athens, Greece
- South Korea (7):
  - GSK Investigational Site, Daegu
  - GSK Investigational Site, Hwasun
  - GSK Investigational Site, Incheon
  - GSK Investigational Site, Jeonju
  - GSK Investigational Site, Pusan
  - GSK Investigational Site, Seoul
  - GSK Investigational Site, Suwon Kyunggi-do

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD will be made available within 6 months of publishing the results of the primary endpoints, key secondary endpoints and safety data of the study.
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: http://clinicalstudydatarequest.com